CLINICAL TRIAL: NCT02743689
Title: Incidence and Perioperative Risk Factors for Early Intensive Care Delirium Following Cardiac Surgery
Brief Title: Perioperative Risk Factors for Intensive Care Delirium After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Vilma Kuzminskaite, MD, Vilnius University
Other Study IDs: DELI-1
Record Dates: First submitted 2016-04-13; First posted 2016-04-19 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Delirium
Keywords: Postoperative; Cardiac surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to identify the incidence of early postoperative delirium in intensive care patients after cardiac surgery and detect possible risk factors associated with increased risk for developing delirium after cardiac surgery.

DETAILED DESCRIPTION:
A consecutive series of patients scheduled for elective cardiac surgery is included in the study. Delirium screening is performed using Intensive Care Delirium Screening Checklist. Preoperative cognitive state is evaluated with Mini-Mental State Examination. Information of possible risk factors is collected from patient's history and chart. The Snoring, Tiredness, Observed apnea, high blood Pressure-Body mass index (BMI), Age, Neck circumference and Gender questionnaire (STOP-BANG questionnaire) is used for obstructive sleep apnea screening.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery
* patient spends more than 1 day in the intensive care unit after the surgery

Exclusion Criteria:

* refusal to participating in the study
* documented severe central nervous system, cognitive or psychiatric disorder
* unable to be screened with Intensive Care Delirium Screening Checklist up to 6th postoperative day (e.g. deeply sedated, intubated patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients scheduled for elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of early postoperative delirium in intensive care patients after cardiac surgery | Within 5 days after the surgery

SECONDARY OUTCOMES:
Perioperative risk factors for delirium after cardiac surgery | Up to 5 postoperative days or occurence of delirium if it develops earlier
  Preoperative risk factors include demographic data, comorbidities and standard preoperative laboratory and instrumental testing results as well as preoperative cognitive status evaluation, performed a day before the surgery. If the patient does not develop delirium, information on intraoperative and postoperative risk factors is collected up to discharge from intensive care unit or maximum 5 postoperative days, whichever happens earlier. If delirium occurs, data on risk factors is collected up to the beginning of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Kuzminskaite, MD, Principal Investigator — Vilnius University Hospital Santariskiu Clinics
Locations (1):
- Vilnius University Hospital Santariskiu Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No